CLINICAL TRIAL: NCT04276649
Title: A Retrospective Analysis on the Influence of Caltrate Supplement on the Clinical Effect of Mesalazine in Ulcerative Colitis
Brief Title: A Retrospective Analysis: the Influence of Caltrate Supplement on the Effect of Mesalazine in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2020-01-103
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis; Vitamin D Deficiency; Vitamin D Supplement
MeSH Terms: conditions — Colitis, Ulcerative; Vitamin D Deficiency | interventions — Calcium Carbonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caltrate+Mesalazine: Patients in this group were received with Caltrate 0.6 g/d and Mesalazine 4g/d orally at least 12 months.
  Interventions: Drug: Caltrate
- Mesalazine: Patients in this group were received with Mesalazine 4g/d orally at least 12 months.

INTERVENTIONS:
Drug: Caltrate — Patients in supplementary group were received with Caltrate 0.6 g/d and Mesalazine 4g/d orally at least 12 months, and those in non-supplementary only take Mesalazine 4g/d.
  Groups: Caltrate+Mesalazine

SUMMARY:
Aims:Retrospectively observe the effects of Caltrate supplementation on the clinical effect of mesalazine in patients with ulcerative colitis.

Design: From January 2015 to December 2020, through retrieving the clinical database of the Second Affiliated Hospital of Wenzhou Medical University, patients with active UC who accepted mesalazine treatment were enrolled. According to whether Caltrate was supplemented at the same time, the patients were divided into supplementary group and non-supplementary group. The modified Mayo score and several laboratory indicators were compared between the two groups.

DETAILED DESCRIPTION:
1. The research has been approved by the Medical Ethics Committee of the Second Affiliated Hospital of Wenzhou Medical University.
2. According to the "Consensus on Diagnosis and Treatment of Inflammatory Bowel Disease" formulated by the Beijing Conference in 2018 as a standard, patients with clear diagnosis of UC are collected. Exclusion criteria included: history of vitamin D treatment within the previous 3 months; treated with glucocorticoids, immunosuppressants, biologic agents, or colectomy during the follow-up; severe liver and kidney dysfunction; other autoimmune diseases.
3. Assess disease activity of UC participants based on the "Mayo score".
4. General information about participants with UC is collected.
5. Serum C-reactive protein, erythrocyte sedimentation rate, white blood cells, albumin, creatinine, calcium and phosphorus levels are measured.
6. The level of serum 25 (OH) D of participants is detected.
7. Participants are divided into two groups, one group was given oral Caltrate 0.6g/d +Mesalazine, and the other group only took Mesalazine .
8. The above serum indicators are re-measured in the 12th month, and the condition of UC participants is also evaluated.
9. Follow-up for 12 months. By comparing the above indicators, observe that in the Han population:

   1. Can Caltrate supplementation increase serum 25 (OH) D levels in patients with UC?
   2. Can Caltrate supplementation improve the condition of patients with UC?
   3. Whether Caltrate works synergistically with Mesalazine?
   4. whether the effect of Caltrate on UC patients is affected by factors such as disease site, disease activity, treatment, etc ..
10. Through statistical analysis, comprehensive analysis of the effectiveness and safety of Caltrate supplementation in Han patients with UC, providing a theoretical basis for further "precise treatment" intervention in inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Clearly diagnosed patients with UC
* Took mesalazine for at least 12 months

Exclusion Criteria:

* had recent supplementation of vitD3
* had prior or concomitant use of other biologic agent, glucocorticoid and/or immunomodulators at the time of enrollment or follow up
* Co-morbid with other autoimmune diseases
* Severe liver and kidney dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Serum 25 (OH) D level | 12 months
  Because serum 25 (OH) D levels are relatively stable, they are considered the most reliable indicator of vitamin D status.
Mayo score | 12 months

SECONDARY OUTCOMES:
erythrocyte sedimentation rate | 12 months
  ESR can be used to reflect the degree of inflammation in the body.
C-reactive protein | 12 months
  C-reactive protein can be used to reflect the degree of inflammation in the human body

CONTACTS AND LOCATIONS:
Overall Officials: Xia sheng long, Master, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- SAHWenzhouMU, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Data sets will be made available on relevant requests and in accordance with journal guidelines when publishing results from this study.